CLINICAL TRIAL: NCT06583811
Title: Remifentanil and Remimazolam to Limit Patient Movement During Long-Eye Surgeries Under Local Anesthesia
Brief Title: Remifentanil and Remimazolam to Limit Patient Movement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Remifentanil and Remimazolam
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-07

CONDITIONS: Long-Eye Surgeries
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Remifentanil Group (Active Comparator): About 35 Patients will receive Remifentanil bolus of 1 μg/kg over 30 seconds followed by a continuous infusion of 0.03-0.05 μg/kg/min.
  Interventions: Drug: Remifentanil
- Group B: Remimazolam Group (Active Comparator): About 35 Patients will receive remimazolam bolus of 0.2mg/kg followed by a continuous infusion of 0.3-0.5 μg/kg/h.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — to compare remifentanil and remimazolam to limit patient movement during long-eye surgeries under local anesthesia.
  Other Names: emimazolam

SUMMARY:
Local anesthetics (LA) may be administered by injection (retrobulbar, peribulbar, subconjunctival, lid, or facial block) or by instillation (topical anesthesia), Considerable drawbacks of local anesthesia in these patients include the fact that a few patients can remain comfortable on an operating table for procedures that exceed two or three hours.

Sedation may be helpful with LA to decrease the experience of discomfort, movement and anxiety, which may in turn positively influence hemodynamic parameters, patient satisfaction, and overall improve surgical safety. Sedatives used in eye surgeries include benzodiazepines, opioids, alpha-adrenoceptor agonists, and propofol.

DETAILED DESCRIPTION:
Ophthalmic surgery is a precise surgical procedure that requires absolute immobilization. Many ophthalmic procedures can be performed safely in an outpatient setting, using local anesthesia.

Propofol is currently the most commonly used intravenous anesthetic. It has a rapid onset of action, a short half-life and is associated with rapid recovery of cognitive ability. However, propofol can lead to injection pain, propofol infusion syndrome, and hemodynamic and respiratory depression. Therefore, there is a need for new anesthetic drugs with high efficacy and fewer side effects while providing stable and controllable anesthesia.

Remifentanil is a short-acting esterase metabolized opioid with analgesic and sedative effects. Its half-life is about 5-10 min so that it can be titrated closely in response to changes in intraoperative requirements and with a low risk of accumulation.

Remimazolam is a novel ultrashort-acting benzodiazepine agonist that works on γ-aminobutyric acid type A (GABA-A) receptors to reduce neuronal excitation and thereby achieve hypoactivity and sedation in the body. Remimazolam is metabolized by a nonspecific esterase, and the metabolite has no pharmacological effect, which allows prolonged infusion without accumulation.

It provides rapid anesthesia and arousal while stabilizing hemodynamics and produces less depression of respiration, making it more suitable for use in elderly and hemodynamically unstable patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Undergoing long-eye surgeries under local anesthesia using peribulbar block with an expected surgical time of more than one hour.

Exclusion Criteria:

* Patients on aspirin or anticoagulants.
* Allergy to any study medication.
* Drug abuse.
* Uncontrolled hypertension.
* Hyperthyroidism.
* Frequent cough.
* Impaired hearing.
* Severe liver and kidney dysfunction.
* Neurological or psychological disorders.
* Partial or failed block.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Eye Movement | from 0 hours to 4 hours after the procedure
  Incidence of patients who are not moving their Eyes during long eye surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided